CLINICAL TRIAL: NCT04212416
Title: A Safety and Feasibility Trial of Leflunomide in Patients With Steroid Dependent Chronic Graft-Versus-Host Disease
Brief Title: Leflunomide in Treating Patients With Steroid Dependent Chronic Graft Versus Host Disease
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19202; NCI-2019-04532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19202 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2019-07-17; First posted 2019-12-27 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Chronic Graft Versus Host Disease; Steroid Refractory Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (leflunomide) (Experimental): Patients receive leflunomide PO QD for days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may optionally continue leflunomide for an additional 6 cycles as long as response or stable disease is maintained.
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — Given PO
  Other Names: Arava; SU101

SUMMARY:
This phase I trial studies the side effects of leflunomide in treating patients with steroid dependent chronic graft versus host disease (cGVHD). cGVHD is a common complication of bone marrow transplant. GVHD occurs when immune cells transplanted from a donor (the graft) recognize the transplant recipient (the host) as foreign, and cause damage to the skin, gastrointestinal tract or other organs. Steroids are the first line of therapy and benefits are seen in about one-third of patients with cGVHD. Prolonged use of steroids is associated with multiple complications. Leflunomide may decrease the body's immune response and reduce inflammation associated with cGVHD.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate safety and tolerability of leflunomide in hematopoietic cell transplant (HCT) patients with steroid dependent chronic GvHD (cGvHD).

SECONDARY OBJECTIVES:

I. Characterize the toxicity profile of leflunomide in patients with steroid dependent cGVHD.

II. Obtain preliminary evidence of leflunomide activity against GVHD by estimating the response rate (as defined by 2014 National Institutes of Health [NIH] consensus development project on clinical trials in cGVHD) in an expansion cohort of 12 patients with steroid dependent cGVHD.

III. Evaluate changes in cGVHD severity using physician-reported cGVHD activity assessment form.

IV. Evaluate changes in symptom activity using cGVHD activity assessment patient self-report.

V. Evaluate failure-free survival and GVHD free survival. VI. Evaluate changes in steroid doses while on therapy. VII. Evaluate rate of infectious complications during leflunomide administration.

EXPLORATORY OBJECTIVES:

I. Assess the presence and percentage of immune cell subsets (including but not limited to Th17 and Treg cells) in whole blood after leflunomide administration.

II. Assess the changes in the presence and levels of GVHD inflammatory biomarkers and cytokines (including but not limited to IL-17A, IL-21, and IL-2) in plasma after leflunomide administration.

III. Assess the plasma pharmacokinetics of teriflunomide (active metabolite of leflunomide).

OUTLINE:

Patients receive leflunomide orally (PO) once daily (QD) for days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may optionally continue leflunomide for an additional 6 cycles as long as response or stable disease is maintained.

After completion of study treatment, patients are followed up at 30 days, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines.
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies.

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval.
* Karnofsky performance status of >= 70 %.
* Ability to read and understand English or Spanish for questionnaires.
* Recipients of allogeneic stem cell transplantation (sibling/unrelated/umbilical cord blood [UCB]/Haplo) with myeloablative or non-myeloablative conditioning regimens.
* Participants must have steroid-dependent cGVHD. Steroid dependent cGVHD is defined as having persistent signs and symptoms of cGVHD despite the use of prednisone for 2 months without complete resolution of signs and symptoms. Both classic cGVHD and overlap syndromes will be allowed to participate.
* Estimated life expectancy greater than 3 months.
* No more than 4 prior lines of treatment. Sirolimus and tacrolimus used for prophylaxis will not be counted as line of therapy.
* Stable dose of corticosteroids for 2 weeks prior to enrollment.
* Able to swallow pills.
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (without myeloid growth factors within 1 week of study entry) (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Platelets >= 50,000/mm^3 (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement.
* Total bilirubin =< 2 mg/dl (exception permitted in patients with Gilbert's syndrome; aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2 x upper limit of normal [ULN]), unless hepatic dysfunction is a manifestation of presumed cGVHD (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).

  * Abnormal liver function tests (LFTs) (liver function panel) in the context of active cGVHD involving other organ systems may also be permitted if the treating physician documents the abnormal LFTs as being consistent with hepatic cGVHD and a liver biopsy will not be mandated in this situation.
* AST =< 2.0 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* ALT =< 2.0 x ULN (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Creatinine clearance of >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal. or calculated by Cockcroft-Gault equation (performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV)*, active hepatitis B virus (HBV) (surface antigen negative), and syphilis (rapid plasma reagin [RPR]) (performed within 28 days prior to day 1 of protocol therapy).

  * If positive, hepatitis C ribonucleic acid (RNA) quantitation must be performed.
* Meets other institutional and federal requirements for infectious disease titer requirements (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).

  * Note: Infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy.
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (to be performed within 28 days prior to day 1 of protocol therapy unless otherwise stated).

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy. The effects of study treatment on a developing fetus have the potential for teratogenic or abortifacient effects. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only).

Exclusion Criteria:

* Exposure to any new immunosuppressive medication in the 4 weeks prior to enrollment.
* Donor lymphocyte infusion within 100 days prior to enrollment.
* Patients may not be receiving any other investigational agents concurrently. Oral chemotherapeutic agents or biologics -for example ruxolitinib or rituximab therapy and ibrutinib / imatinib (either past or current exposure) - is allowed.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent.
* Active infection requiring antibiotics. An active uncontrolled infection is defined as hemodynamic instability attributed to sepsis or new symptoms, worsening physical signs, or radiographic findings attributable to infection. Persisting fever without signs or symptoms will not be interpreted as an active uncontrolled infection.
* Uncontrolled cardiac angina or symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV).
* Pregnant women are excluded from this study. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with leflunomide.
* Patients should not have any uncontrolled illness including ongoing or active infection.
* Active malignant relapse.
* Patients with other active malignancies are ineligible for this study, other than superficial localized skin cancer (basal or squamous cell carcinoma).
* Active diarrhea, not related to cGVHD.
* Clinically significant uncontrolled illness.
* Patients on dialysis.
* Patients requiring ventilator support.
* Patients with acute GvHD
* Known history of immunodeficiency virus (HIV) or hepatitis B or hepatitis C infection.
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
* Inability to comply with protocol therapy and follow up visits.
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2026-06-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity | Up to 28 days
  Toxicity will be graded according to the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v.5.0).

SECONDARY OUTCOMES:
Leflunomide activity | At 24 weeks
  Leflunomide activity in patients with steroid dependent chronic graft versus host disease (cGVHD) and disease status at 24 weeks in terms of partial and complete response will be evaluated as defined by 2014 National Institutes of Health (NIH) consensus development project on clinical trials in cGVHD.
Changes in cGVHD severity | Baseline up to 30 days post treatment
  Evaluated using physicians-reported cGVHD activity assessment form.
Changes in symptom activity | Baseline up to 30 days post treatment
  Evaluated using cGVHD activity assessment patient self-report.
Failure-free survival | At 24 weeks
  Defined by the absence of second line of GVHD treatment, non-relapse mortality, and recurrent malignancy during leflunomide treatment. Failure free survival estimates will be calculated using the Kaplan-Meier method.
Failure-free survival | At 28 days follow-up
  Defined by the absence of second line of GVHD treatment, non-relapse mortality, and recurrent malignancy during leflunomide treatment. Failure free survival estimates will be calculated using the Kaplan-Meier method.
GVHD-free survival | At 24 weeks
  Defined as the probability of being alive without clinically significant GvHD at any time-point post transplantation.
GVHD-free survival | At 28 days follow-up
  Defined as the probability of being alive without clinically significant GvHD at any time-point post transplantation.
Changes in steroid doses while on therapy | Baseline up to 48 weeks
  Will be recorded and assessed at each study visit time-points.
Rate of infectious complications | Up to 48 weeks
  Will be evaluated while on therapy.

OTHER OUTCOMES:
Presence and levels of immune cells (i.e., T and B cells, regulatory T cells [T regs], T cell receptor excision circles [TRECs]) after leflunomide consumption | Up to 28 days follow-up
  Will be determined using flow cytometric analysis on freshly thawed peripheral blood mononuclear cells (PBMNCs).
Effect of leflunomide consumption of the presence and levels of GVHD inflammatory biomarkers | Up to 48 weeks
  Will be assessed by performing enzyme-linked immunosorbent assay (ELISA) assays on freshly thawed serum samples.
Pharmacokinetics concentration of teriflunomide in patients with chronic GVHD | Up to 28 days follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Amandeep Salhotra, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States